CLINICAL TRIAL: NCT00698841
Title: A Study to Evaluate the Relationship Between Cetuximab Therapy and Corrected QT (QTc) Interval Changes in Patients With Advanced Malignancies From Solid Tumors
Brief Title: Study to Evaluate the Effect of Cetuximab on Corrected QT (QTc) Interval Changes in Patients With Advanced Malignancies From Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-315
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Results first posted 2011-05-11 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab (Experimental)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab administered by intravenous (IV) infusion at an initial dose of 400 mg/m^2 over 120 minutes on Day 1 followed by a weekly maintenance IV dose of 250 mg/m^2 over 60 minutes.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to determine whether corrected QT (QTc) interval changes occur on an electrocardiogram (ECG) when cetuximab is administered to the study population.

ELIGIBILITY:
Inclusion criteria:

* Advanced or metastatic malignant disease originating from solid tumors
* Adequate recovery from previous therapy or intervention; at least 21 days since major surgery or prior radiation therapy
* Measurable or evaluable disease

Exclusion criteria:

* Women of childbearing potential (WOCBP) who are breastfeeding, pregnant, or unwilling or unable to use acceptable contraception during the study and for at least 12 weeks after the last on-study dose of cetuximab
* Men unwilling to use acceptable contraception during the study if engaged in sexual relations with a WOCBP
* Symptomatic brain metastasis
* History of myocardial infarction 6 months or less prior to study entry, of severe congestive heart failure, of uncontrolled angina, or of uncontrolled arrhythmias
* Clinically relevant abnormality on screening electrocardiogram (ECG), preventing an accurate measurement of the QT interval
* Congenital long QT syndrome
* History of risk factors for ventricular tachycardia or Torsades de pointes or history of fainting, unexplained loss of consciousness, or convulsions
* Prolonged QTc interval on screening ECG (greater than 470 msec) using Fridericia's correction formula
* Heart rate slower than 50 bpm or faster than 100 bpm at rest during screening ECG measurements
* Implantable pacemaker or automatic implantable cardioverter defibrillator
* Sustained supine systolic blood pressure higher than 150 mmHg or lower than 90 mmHg or a diastolic blood pressure lower than 45 mmHg or higher than 95 mmHg at screening
* Known history of arterial thrombotic events within 6 months prior to study initiation
* Known history of significant peripheral artery disease
* Current participation in a clinical trial with another investigational new drug or device
* Receipt of an investigational new drug or device within 21 days prior to enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- United States (15):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Donald W. Hill, MD, Casa Grande, Arizona
  - Compassionate Cancer Care Medical Group, Inc, Corona, California
  - Compassionate Cancer Care Medical Group Inc, Fountain Valley, California
  - Pacific Shores Medical Group, Long Beach, California
  - Desert Hospital Comprehensive Cancer Center, Palm Springs, California
  - Compassionate Cancer Care Medical Group, Inc, Riverside, California
  - American Institute Research, Whittier, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Baptist Cancer Institute, Jacksonville, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Brinz, Burroff, Gurtler, & Russo, Metairie, Louisiana
  - Cancer Specialists Of Oklahoma, Oklahoma City, Oklahoma
  - Pharma Resource, East Providence, Rhode Island
  - Austin Cancer Centers, Austin, Texas
- Local Institution, San Juan, Pr, Puerto Rico

REFERENCES:
- [Derived] Deeken JF, Shimkus B, Liem A, Hill D, Gurtler J, Berghorn E, Townes L, Lu H, Trifan O, Zhang S. Evaluation of the relationship between cetuximab therapy and corrected QT interval changes in patients with advanced malignancies from solid tumors. Cancer Chemother Pharmacol. 2013 Jun;71(6):1473-83. doi: 10.1007/s00280-013-2146-5. Epub 2013 Apr 16. PMID 23589315
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 79 participants enrolled, 51 received treatment.
Groups:
- Cetuximab: Cetuximab given by intravenous (IV) infusion at an initial dose of 400 mg/m^2 over 120 minutes on Day 1 followed by a weekly maintenance IV dose of 250 mg/m^2 over 60 minutes.
Period: Overall Study
Arm/Group | Cetuximab
Started | 51
Completed | 33
Not Completed | 18
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 3
Not completed — Disease progression | 7
Not completed — Failure to meet eligibility criteria | 2
Not completed — Study drug toxicity | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 45
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Meaningful Prolongation of the QT Interval Corrected for Heart Rate (QTc) From Time-matched Baseline
Description: 12-Lead continuous digital electrocardiogram (ECG) data were collected at preselected time points at baseline visit and on Days 1, 8, 15, 22, and 29. The QT interval is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. The corrected QTc is the QT interval corrected for heart rate. Prolongation of the QTc was identified as clinically meaningful at the investigator's discretion.
Time Frame: Baseline, Day 1, and then weekly to end of Cycle 1 (28 days)
Population: Those who met all study criteria and did not require interrupted cetuximab infusion on Day (D)1 or 22; miss an ECG timepoint at baseline, D1, or D22; stop/modify dose of a scheduled drug that prolongs QT/QTc interval, receive other cancer therapy, begin a prohibited drug, or require cetuximab dose reduction before D29; withdraw consent before D23.
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 37
Participants | 0

2. Secondary Outcome: Number of Participants With Clinically Significant Changes in PR Interval, QRS Interval, and Heart Rate
Description: 12-Lead continuous digital ECG data were collected at preselected time points at baseline visit and on Days 1, 8, 15, 22, and 29. The PR interval is the time from the onset of the P wave to the beginning of the QRS complex. The QRS interval=deflections in the ECG, comprising Q, R, and S waves, that represent depolarization of the ventricles. Clinically significant was determined at the investigator's discretion.
Time Frame: Baseline, Day 1, and then weekly to end of Cycle 1 (28 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 37
Participants
  Changes in PR interval | 0
  Changes in QRS interval | 0
  Changes in heart rate | 0

3. Secondary Outcome: Number of Participants With Death, Treatment-related Death, Serious Adverse Events (SAEs), Treatment-related SAEs, Adverse Events (AEs) Leading to Discontinuation, and Treatment-related AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with treatment. SAE=any untoward medical occurrence that at any dose results in death, is life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, or is an important medical event. Treatment related=possibly, probably, or certainly related to or of unknown relationship to study treatment.
Time Frame: Baseline through Cycle 1 (28 days), continuously
Population: All participants who received at least 1 dose of cetuximab.
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 51
Participants
  Deaths | 6
  Treatment-related deaths | 0
  SAEs | 16
  Treatment-related SAEs | 2
  AEs leading to discontinuation | 10
  Treatment-related AEs leading to discontinuation | 3

4. Secondary Outcome: Number of Participants With AEs of Special Interest by Worst Common Terminology Criteria (CTC) Grade
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with treatment. AEs of special interest have been sponsor-selected based on the known clinical effects of cetuximab. Treatment related=possibly, probably, or certainly related to or of unknown relationship to study treatment. CTC Grade 1: Mild. Grade 2: Moderate. Grade 3: Severe or medically significant but not immediately life-threatening. Grade 4: Life-threatening.
Time Frame: Baseline through Cycle 1 (28 days), continuously
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 51
Participants
  Infusion reaction (Any grade) | 6
  Infusion reaction (Grade 3) | 2
  Infusion reaction (Grade 4 or 5) | 0
  Acneform rash (Any grade) | 32
  Acneform rash (Grade 3) | 1
  Acneform rash (Grade 4 or 5) | 0
  Cardiac event (Any grade) | 2
  Cardiac event (Grade 3) | 1
  Cardiac event (Grade 4 or 5) | 0
  Treatment-related infusion reaction (Any grade) | 6
  Treatment-related infusion reaction (Grade 3) | 2
  Treatment-related infusion reaction (Grade 4 or 5) | 0
  Treatment-related acneform rash (Any grade) | 31
  Treatment-related acneform rash (Grade 3) | 1
  Treatment-related acneform rash (Grade 4 or 5) | 0
  Treatment-related cardiac event (Any grade) | 0
  Treatment-related cardiac event (Grade 3) | 0
  Treatment-related cardiac event (Grade 4 or 5) | 0

5. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities by Worst CTC Grade at Baseline and On-study
Description: BL=baseline; OS=on-study; ULN=upper level of normal. Albumin,low (g/dL) Grade 1:<LLN-30, Grade 2:<30-20, Grades 3&4:<20. Aspartate aminotransferase (AST)(U/L) Grade 1:>ULN-2.5*ULN, Grade 2:>2.5-5.0*ULN, Grade 3:>5.0-20.0*ULN, Grade 4:>20.0*ULN. Total bilirubin, high Grade 1:ULN-1.5*ULN, Grade 2:>1.5-3.0*ULN, Grade 3:>3.0-10.0*ULN, Grade 4:>10.0*ULN. Alkaline phosphatase (ALP) (U/L) Grade 1:>ULN-2.5*ULN, Grade 2:>2.5-5.0*ULN, Grade 3:>5.0-20.0*ULN, Grade 4:>20.0*ULN. Creatinine (mg/dL) Grade 1:>ULN-1.5*ULN, Grade 2:>1.5-3.0*ULN, Grade 3:>3.0-6.0*ULN, Grade 4:>6.0*ULN.
Time Frame: At screening, at the end of Cycle 1 (28 days)
Population: All participants who received at least 1 dose of cetuximab
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 51
Participants
  Albumin, low (BL, Grades 1-4) ( N=48) | 18
  Albumin, low (OS, Grade 1-4) ( N=45) | 27
  Albumin, low (BL, Grades 3 or 4) ( N=48) | 0
  Albumin, low (OS, Grades 3 or 4) ( N=45) | 0
  Albumin, low (BL, Grade 4) (N=48) | 0
  Albumin, low (OS, Grade 4) (N=45) | 0
  AST, high (BL, Grades 1-4) ( N=48) | 9
  AST, high (OS, Grades 1- 4) ( N=45) | 19
  AST, high (BL, Grades 3 or 4) ( N=48) | 1
  AST, high (OS, Grades 3 or 4) ( N=45) | 2
  AST, high (BL, Grade 4) ( N=48) | 0
  AST, high (OS, Grade 4) ( N=45) | 0
  Total bilirubin, high (BL, Grades 1-4) ( N=48) | 2
  Total bilirubin, high (OS, Grades 1-4) ( N=45) | 4
  Total bilirubin, high (BL, Grades 3 or 4) ( N=48) | 0
  Total bilirubin, high (OS, Grades 3 or 4) (N=45) | 1
  Total bilirubin, high (BL, Grade 4) ( N=48) | 0
  Total bilirubin, high (OS, Grade 4) ( N=45) | 0
  ALP, high (BL, Grade 1-4) ( N=48) | 18
  ALP, high (OS, Grade 1-4) ( N=45) | 25
  ALP, high (BL, Grade 3 or 4) ( N=48) | 1
  ALP, high (OS, Grade 3 or 4) ( N=45) | 2
  ALP, high (BL, Grade 4) ( N=48) | 0
  ALP, high (OS, Grade 4) ( N=45) | 0
  Creatinine, high (BL, Grades 1-4) ( N=48) | 1
  Creatinine, high (OS, Grade 1-4) ( N=45) | 2
  Creatinine, high (BL, Grades 3 or 4) ( N=48) | 0
  Creatinine, high (OS, Grades 3 or 4) ( N=45) | 0
  Creatinine, high (BL, Grade 4) ( N=48) | 0
  Creatinine, high (OS, Grade 4) ( N=45) | 0

6. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities by Worst CTC Grade at Baseline and On-study (Continued)
Description: BL=baseline; OS=on-study; LLN=lower level of normal; ULN=upper level of normal. Sodium, low(mmol/L) Grades 1&2:<LLN-130, Grade 3:<130-120, Grade 4:<120. Sodium, high (mmol/L) Grade 1:>ULN-150, Grade 2:>150-155, Grade 3:>155-160, Grade 4:>160. Potassium, high (mmol/L) Grade 1:>ULN-5.5, Grade 2:>5.5-6.0, Grade 3:>6.0-7.0, Grade 4:>7.0. Glucose, low(mg/dL) Grade 1:<LLN-55, Grade 2:<55-40, Grade 3:<40-30, Grade 4:<30. Glucose, high (mg/dL) Grade 1:>ULN-160, Grade 2:>160-250, Grade 3:>250-500, Grade 4:>500. Calcium, high(mg/dL) Grade 1:>ULN-11.5, Grade 2:>11.5-12.5, Grade 3:>12.5-13.5, Grade 4:>13.
Time Frame: At screening, at the end of Cycle 1 (28 days)
Population: All participants who received at least 1 dose of cetuximab
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 51
Participants
  Sodium, low (BL, Grades 1-4) ( N=48) | 0
  Sodium, low (OS, Grades 1- 4) ( N=45) | 7
  Sodium, low (BL, Grades 3 or 4) ( N=48) | 15
  Sodium, low (OS, Grades 3 or 4) ( N=45) | 2
  Sodium, low (BL, Grade 4) ( N=48) | 0
  Sodium, low (OS, Grade 4) ( N=45) | 0
  Sodium, high (BL, Grade 1-4) ( N=48) | 1
  Sodium, high (OS, Grades 1-4) ( N=45) | 5
  Sodium, high (BL, Grades 3 or 4) ( N=48) | 0
  Sodium, high (OS, Grades 3 or 4) ( N=45) | 0
  Sodium, high (BL, Grade 4) ( N=48) | 0
  Sodium, high (OS, Grade 4) ( N=45) | 0
  Potassium, high (BL, Grades 1-4) ( N=48) | 2
  Potassium, high (OS, Grades 1-4) ( N=45) | 3
  Potassium, high (BL, Grade 3 or 4) ( N=48) | 0
  Potassium, high (OS, Grade 3 or 4) ( N=45) | 1
  Potassium, high (BL, Grade 4) ( N=48) | 0
  Potassium, high (OS, Grade 4) ( N=45) | 0
  Glucose, low (BL, Grades 1- 4) ( N=48) | 0
  Glucose, low (OS, Grades 1-4) ( N=45) | 2
  Glucose, low (BL, Grades 3 or 4) ( N=48) | 0
  Glucose, low (OS, Grades 3 or 4) ( N=45) | 0
  Glucose, low (BL, Grade 4) ( N=48) | 0
  Glucose, low (OS, Grade 4) ( N=45) | 0
  Glucose, high (BL, Grades 1- 4) ( N=48) | 29
  Glucose, high (OS, Grades 1- 4) ( N=45) | 37
  Glucose, high (BL, Grades 3 or 4) (N=48) | 2
  Glucose, high (OS, Grades 3 or 4) (N=45) | 4
  Glucose, high (BL, Grade 4) (N=48) | 0
  Glucose, high (OS, Grade 4) (N=45) | 0
  Calcium, low (BL, Grade 1-4) (N=48) | 4
  Calcium, low (OS, Grade 1-4) (N=45) | 14
  Calcium, low (BL, Grade 3 or 4) (N=48) | 0
  Calcium, low (OS, Grades 3 or 4) (N=45) | 0
  Calcium, low (BL, Grade 4) (N=48) | 0
  Calcium, low (OS, Grade 4) (N=45) | 0
  Calcium, high (BL, Grades 1-4) (N=48) | 2
  Calcium, high (OS, Grades 1-4) (N=45) | 2
  Calcium, high (BL, Grades 3 or 4) (N=48) | 0
  Calcium, high (OS, Grades 3 or 4) (N=45) | 0
  Calcium, high (BL, Grade 4) (N=48) | 0
  Calcium, high (OS, Grade 4) (N=45) | 0
  Magnesium, low (BL, Grades 1-4) (N=41) | 3
  Magnesium, low (OS, Grades 1-4) (N=38) | 11
  Magnesium, low (BL, Grades 3 or 4) (N=41) | 0
  Magnesium, low (OS, Grades 3 or 4) (N=38) | 1
  Magnesium, low (BL, Grade 4) (N=41) | 0
  Magnesium, low (OS, Grade 4) (N=38) | 1

7. Primary Outcome: Mean Change in QTc From Time-matched Baseline Assessed Using Fridericia's Correction Formula (QTcF) by Study Day and Time Point
Description: The QT interval is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. The QTc is the QT interval corrected for heart rate. The QTcF=QT/RR^1/3, where RR=RR interval in seconds. Baseline=predose. Mean change in QTc interval from baseline to time t=QTc interval at time t minus QTc interval at baseline.
Time Frame: Predose Day 1 (Baseline) to end of Cycle 1 (28 days)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Cetuximab
Number analyzed (Participants) | 37
msec
  Day 1 (N=36) Predose | 3.8 (2.5)
  Day 1 (N=37) 1 hour | 1.8 (1.9)
  Day 1 (N=37) 2 hour | 0.7 (2.1)
  Day 1 (N=36) 3 hour | 1.2 (1.6)
  Day 1 (N=37) 6 hour | -2.4 (1.8)
  Day 8 (N=37) Predose | 1.3 (2.2)
  Day 8 (N=37) 1 hour | 1.9 (2.5)
  Day 8 (N=37) 2 hour | 4.5 (2.7)
  Day 8 (N=36) 3 hour | 0.8 (2.5)
  Day 15 (N=37) Predose | 3.2 (2.7)
  Day 15 (N=37) 1 hour | 2.6 (3.1)
  Day 15 (N=37) 2 hour | 1.2 (3.2)
  Day 15 (N=36) 3 hour | -0.7 (3.6)
  Day 22 (N=37) Predose | 2.3 (3.3)
  Day 22 (N=37) 1 hour | 3.4 (2.9)
  Day 22 (N=37) 2 hour | 4.1 (3.2)
  Day 22 (N=36) 3 hour | 2.2 (2.8)
  Day 22 (N=37) 6 hour | 2.6 (2.4)
  Day 29 (N=30) Predose | 0.0 (3.4)
  Day 29 (N=30) 1 hour | 3.5 (2.9)
  Day 29 (N=30) 2 hour | 3.5 (2.7)
  Day 29 (N=29) 3 hour | 4.0 (3.0)

8. Secondary Outcome: Number of Participants With Hematology Abnormalities by Worst CTC Grade at Baseline and On-study
Description: BL=baseline; OS=on-study; LLN=lower level of normal. Laboratory values assessed using CTC for AEs, Version 3.0. Hemoglobin (g/dL) Grade 1:<LLN to 10.0, Grade 2:<10.0 to 8.0, Grade 3:<8.0 to 6.5, Grade 4:<6.5. Platelets Grade 1:LLN to 75.0*10^9/L, Grade 2:<75.0 to 50.0*10^9/L, Grade 3:<50.0 to 25.0*10^9/L, Grade 4:<25.0 to 10^9/L. White blood cells Grade 1:<LLN to 3.0*10^9/L, Grade 2:<3.0 to 2.0*10^9/L, Grade 3:<2.0 to 1.0*10^9/L, Grade 4:<1.0*10^9/L. Neutrophils Grade 1:<LLN to 1.5*10^9/L, Grade 2:<1.5 to 1.0*10^9/L, Grade 3:<1.0 to 0.5*10^9/L, Grade 4:<0.5*10^9/L.
Time Frame: At screening, weekly prior to start of cetuximab infusion, at end of Cycle 1 (28 days), and at 30-day follow-up
Population: All participants who received at least 1 dose of cetuximab.
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 51
Participants
  Hemoglobin, low (BL, Grades 1-4) (N=51) | 35
  Hemoglobin, low (OS, Grades 1-4) (N=45) | 34
  Hemoglobin, low (BL, Grades 3 or 4) (N=51) | 1
  Hemoglobin, low (OS, Grades 3 or 4) (N=45) | 2
  Hemoglobin, low (BL, Grade 4) (N=51) | 0
  Hemoglobin, low (OS, Grade 4) (N=45) | 0
  Platelets, low (BL, Grades 1-4) (N=51) | 8
  Platelets, low (OS, Grades 1-4) (N=45) | 9
  Platelets, low (BL, Grades 3 or 4) (N=51) | 0
  Platelets, low (OS, Grades 3 or 4) (N=45) | 0
  Platelets, low (BL, Grade 4) (N=51) | 0
  Platelets, low (OS, Grade 4) (N=45) | 0
  White blood cells, low (BL, Grades 1-4) (N=51) | 4
  White blood cells, low (OS, Grades 1-4) (N=45) | 13
  White blood cells, low (BL, Grades 3 or 4) (N=51) | 0
  White blood cells, low (OS, Grades 3 or 4) (N=45) | 0
  White blood cells, low (BL, Grade 4) (N=51) | 0
  White blood cells, low (OS, Grade 4) (N=45) | 0
  Neutrophils, low (BL, Grades 1-4) (N=47) | 0
  Neutrophils, low (OS, Grades 1-4) (N=44) | 5
  Neutrophils, low (BL, Grade 3 or 4) (N=47) | 0
  Neutrophils, low (OS, Grade 3 or 4) (N=44) | 1
  Neutrophils, low (BL, Grade 4) (N=47) | 0
  Neutrophils, low (OS, Grade 4) (N=44) | 0

ADVERSE EVENTS:
Time Frame: Baseline through Cycle 1 (28 days) and up to 30 following last dose of study medication (totaling up to 58 days)
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 16/51
Other Adverse Events (participants affected / at risk) | 43/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=51)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
HEADACHE (Nervous system disorders) | 1
ASCITES (Gastrointestinal disorders) | 1
DISTAL INTESTINAL OBSTRUCTION SYNDROME (Gastrointestinal disorders) | 1
SEPSIS (Infections and infestations) | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
PAIN (General disorders) | 1
DISEASE PROGRESSION (General disorders) | 4
INFUSION RELATED REACTION (General disorders) | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NASOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=51)
WEIGHT DECREASED (Investigations) | 3
HEADACHE (Nervous system disorders) | 11
NAUSEA (Gastrointestinal disorders) | 6
VOMITING (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 4
URINARY TRACT INFECTION (Infections and infestations) | 4
ANAEMIA (Blood and lymphatic system disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 22
PRURITUS (Skin and subcutaneous tissue disorders) | 3
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 3
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 9
CHILLS (General disorders) | 3
FATIGUE (General disorders) | 5
PYREXIA (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.